CLINICAL TRIAL: NCT03993067
Title: Hemopatch as a Tool to Prevent Biliary Fistula in Liver Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Director of the Department of Surgery Head of the General and Hepatobiliary surgery unit, Clinical Professor and Principal investigator, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HBF2018
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Biliary Fistula; Surgery
MeSH Terms: conditions — Biliary Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (Active Comparator): Fibrin glue and Tabotamp on cut surface
  Interventions: Procedure: Fribrin glue and Tabotamp
- Hemopatch (Experimental): Hemopatch on cut surface
  Interventions: Procedure: Hemopatch

INTERVENTIONS:
Procedure: Hemopatch — Hemopatch is a collagen based sealant is a hemostat agent. We want to investigate his role in the prevention of post operative biliary fistula
  Other Names: Experimental
  Arms: Hemopatch
Procedure: Fribrin glue and Tabotamp — Fibrin glue and Tabotampis the standard treatment
  Other Names: Standard treatment
  Arms: Standard Treatment

SUMMARY:
The aim of the study is to investigate the use of Hemopatch to prevent biliary fistula in patients submitted to surgery for malignancy.

DETAILED DESCRIPTION:
Background: Biliary fistula (BF) is one of the most common sources of post hepatectomy morbidity. International Study Group of Liver Surgery (ISGLS) define BF as increased bilirubin concentration in the drain at least 3 times greater than the serum bilirubin concentration on or after postoperative day (POD) 3. BF is graded into grade A, B and C, based on the clinical impact on the postoperative course. Considering ISGLS definition, the incidence of BF ranges from 4,4% to 27,2%. The definition developed in Humanitas Research Hospital (HRH), defines BF as bilirubin concentration in the drain fluid greater than 10 mg/dL on or after POD 3. In this case, the incidence is around 8%. Various topical haemostatic agents have been developed for liver resection area management their usefulness in preventing BF by using a sealing product on the resection surface still remains unclear and needs to be assessed.

Objective: this study aimed to assess the clinical validation of Hemopatch to prevent post-operative biliary fistula. Secondarily, it is aimed to evaluate the clinical validity of the two proposed definition of biliary fistula.

Methods: According to the incidence of BF in our previous series (considering ISGLS definition), we designed a randomized controlled study on 220 patients, who underwent hepatic resection from 2018 to 2020. Patients were randomized to treatment group A (Hemopatch) and standard group B (Tisseal and Tabotamp). Both ISGLS and HRH definitions of BF were considered. All patients were systematically drained. Drains were maintained at least 5 days, and bilirubin was measured on PODs 3, 5, and 7. Drains were removed if the bilirubin concentration in the drain fluid was less than 10 mg/dL on POD 7. A statistical analysis to compare perioperative variables between two groups was performed. Then, a multivariate analysis was performed to identify potential risk factors for BF.

ELIGIBILITY:
Inclusion Criteria:

* all patients submitted to liver surgery for malignancies.
* >18 years of age.

Exclusion Criteria:

* biliary reconstruction
* other associated visceral resections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
The rate of biliary fistula | 12 months
  Use a Hemopatch to prevent biliary fistula

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, Principal Investigator — Department of Biomedical Sciences Humanitas University, Milan
Locations (1):
- Department of Hepatobiliary and General Surgery, Humanitas Research Hospital, University of Milan, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No